CLINICAL TRIAL: NCT06709248
Title: Feasibility of a Group-Based Intervention to Enhance Health-Related Quality of Life and Physical Activity in Children and Adolescents With Chronic Illness: A Study Protocol
Brief Title: Feasibility of a Life Coping Program: A Study Protocol
Acronym: LifeCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 578213; Recruitment PhD (Other Grant/Funding Number: University of Bergen, Deparment of Medicine)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-11

CONDITIONS: Health Literacy; Health Related Quality of Life; Physical Activity; Pediatric ALL
MeSH Terms: conditions — Motor Activity; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): In this feasability study following established clinical practice, all participants are included in the intervention Life Coping Program.
  Interventions: Behavioral: Life Coping Program

INTERVENTIONS:
Behavioral: Life Coping Program — The Life Coping Program is built around a coordinated 5-day Life Coping Course. Participants included are grouped by their primary condition, meaning the diagnosis or illness reasoning the referral. Each family is assigned a dedicated Primary Contact throughout the program, and the program consists of three phases: Phase 1: Preparation - Written/visual materials and questionnaires are provided to motivate and inform. A digital consultation occurs 3-5 weeks before the Life Coping Course, covering goals, commitment, and follow-up. Materials are offered in paper or digital formats. Phase 2: Life Coping Course - The 5-day course includes individual consultations, group activities, education, and medical follow-ups, focusing on coping strategies and well-being. Phase 3: Implementation - A summary meeting is conducted, including key persons for further implementation in own local area. Digital follow-ups at 3-4 weeks and 6 months post course assess progress and guide goal achievement.

SUMMARY:
The goal of this observational study is to evaluate the feasibility of the intervention Life Coping Program in children and adolescents 8-16 years of age. The main question it aims to answer is:

Is the Life Coping Program in its current form feasible among children and adolescents with a variety of primary conditions?

The health care providers of participants already undergoing the Life Coping Program will answer survey questions after key procedures of the intervention, and the research team will be given access to measures provided by the participants.

DETAILED DESCRIPTION:
Feasibility and acceptability of the intervention Life Coping Program will be evaluated in an uncontrolled open-label trial using quantitative measures. Sixty children or adolescents with chronic illness or severe medical condition will be recruited along with one associated caregiver. Feasibility will be assessed by tracking attendance and participation in different parts of the intervention. Acceptability of the intervention will be assessed using patient reported experience measures (PREM). Health related quality of life (HrQoL) and level of physical activity will be measured using the Kidscreen 27 and Actigraph GT3X+ monitor, respectively, at baseline and post-intervention.

The study is based on the British Medical Research Council's (MRC) framework for developing and evaluating complex interventions, and will explore innovative treatment strategies that could potentially improve current clinical outcomes and reduce the need for ongoing healthcare follow-up. The findings from this feasibility study will lay the groundwork for a future definitive randomized controlled trial in accordance with the MRC framework for developing and evaluating complex interventions.

ELIGIBILITY:
Inclusion Criteria:

* Have received treatment at Haukeland University Hospital
* One or more of the following primary conditions: congenital heart defects, congenital oral clefts, premature birth before 32 weeks of gestation, completion of cancer treatment, chronic pain conditions, or significant burn injuries
* Must be able to answer questionnaires in Norwegian

Exclusion Criteria:

* Medical condition that may hinder og alter participation
* Treatment plan that may hinder or alter participation

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of completed components | From enrollment to 6 months after the 5-day Life Coping Course
  The proportion of completed components of the Life Coping Program per participant, as reported on checklists completed by health personnel, fully completed questionnaires by participants, and successful use of activity monitors.
Checklist for health personnel | Immediately after the procedures
  Based on the work of Bellg et al. (2004) and Husted et al. (2014), purpose-built checklists are designed for four pre-defined key procedures of the intervention;
  1. Primary digital consultation,
  2. primary individual consultation during the Life Coping Course,
  3. Activities during the Life Coping Course, and
  4. The digital follow-up consultation 3-4 weeks after.

SECONDARY OUTCOMES:
Evaluation of the Life Coping Course | Immediately after the procedure
  A purpose-design evaluation form aiming to assess adolescent and caregivers' experiences and acceptance of phase 2: the five-day Life Coping Course. The questionnaire covers practical aspects, perceived relevance of the activities, interactions with healthcare staff, and overall alignment with their life situation
Health related Quality of Life | From enrollment to 3-4 weeks and 6 months after the 5-days Life Coping Course
  The standardised and valid questionnaire KidScreen27 will be used. Both the version for children and adolescents and the version for parents will be implemented in the study.
Activity Levels | From enrollment to 6 months after the 5-days Life Coping Course
  Objective activity levels will be measured using ActiGraph GT3X+-monitors following a standardized protocol of seven consecutive days of measuring.
Self-reported activity levels and satisfaction with relevant activities | From enrollment to 3-4 weeks and 6 months after the five-day Life Coping Course.
  A purpose-made questionnaire aiming on investigating the child or adolescents relations to physical activity. The questionnaire is partly based on the WHO-survey "Health Behavior in School-Aged Children".

CONTACTS AND LOCATIONS:
Overall Officials: Mette Engan, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland university hospital - Department of Pediatrics, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bovim LPV, Rotevatn EO, Kvidaland HK, Bogen B, Halvorsen T, Engan M. Feasibility of a group-based intervention to enhance health-related quality of life and physical activity in children and adolescents with chronic illness: a study protocol. Pilot Feasibility Stud. 2025 Jul 17;11(1):101. doi: 10.1186/s40814-025-01682-w. PMID 40676648
- See also: (NORWEGIAN) Brief description of the intervention Life Coping Program, as presented to the public — https://www.helse-bergen.no/avdelinger/barne-og-ungdomsklinikken/energisenteret/mestringsuker/
- See also: (NORWEGIAN) Open part of the digital portal — https://app-mestringsukene.youwell.no/prg/p

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT06709248/SAP_000.pdf